CLINICAL TRIAL: NCT01824758
Title: The Effect of Esmolol on Pain Due to Rocuronium Injection Pain
Brief Title: Effect of Esmolol on Pain Due to Rocuronium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, Specialist, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ESM 0538
Record Dates: First submitted 2013-03-01; First posted 2013-04-05 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Injection Site Irritation
Keywords: esmolol, injection pain, lidocaine, rocuronium
MeSH Terms: interventions — Lidocaine; esmolol; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- brevibloc (esmolol) (Experimental): Group E will receive esmolol (1 mg/kg), Group L lidocaine (0.5 mg/kg)and Group C placebo(NaCl 0.9%, 5 mL)
  Interventions: Drug: Esmolol; Drug: rocuronium
- Aritmal (Lidocaine) (Active Comparator): Group E: esmolol (1 mg/kg) Group L: lidocaine (0.5 mg/kg) Group C: placebo(NaCl 0.9%, 5 mL)
  Interventions: Drug: Lidocaine; Drug: rocuronium
- Placebo (NaCl 0.9%, 5 ml) (Placebo Comparator): Group E: esmolol (1 mg/kg) Group L: lidocaine (0.5 mg/kg) Group C: placebo(NaCl 0.9%, 5 mL)
  Interventions: Drug: rocuronium; Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Group L lidocaine (0.5 mg/kg), (rocuronium) (0.05mg/kg).
  Other Names: Aritmal, Jetmonal
  Arms: Aritmal (Lidocaine)
Drug: Esmolol — Group E: esmolol (1 mg/kg), (rocuronium) (0.05mg/kg)
  Other Names: brevibloc
  Arms: brevibloc (esmolol)
Drug: rocuronium — 0.05 mg/kg rocuronium
Drug: Placebo — Group C: Placebo (NaCl 0.9%, 5 ml), (rocuronium) (0.05mg/kg)
  Arms: Placebo (NaCl 0.9%, 5 ml)

SUMMARY:
90 American society of anesthesiology (ASA) physical status I and II patients undergoing general anesthesia for elective surgery will be included in the study. Patients will be randomized into three groups. Group E will receive esmolol (1 mg/kg), Group IL lidocaine (0.5 mg/kg)and Group C placebo(NaCl 0.9%, 5 mL), followed by a 0.05 mg/kg rocuronium. After intravenous induction with propofol, adequate muscle relaxation for intubation will be received by 0.5 mg/kg rocuronium.

DETAILED DESCRIPTION:
Patients will be observed after injection of rocuronium 0.05mg/kg, then immediately asked if they have pain in the arm. The response are assessed; discomfort, pain, and withdrawal of the hand are recorded and graded using a 4-point scale (none, mild, moderate, or severe). After the intubating dose of rocuronium, withdrawal reactions are scored as follows: (a) no pain response, (b)pain limited to the wrist, (c) pain limited to the elbow/shoulder, or (d) generalized pain response.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II patients
* Undergoing general anesthesia for elective surgery

Exclusion Criteria:

* Known allergy to esmolol or lidocaine
* Chronic pain
* Pregnancy
* Withdrawal of consent by the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The injection pain due to rocuronium | 1 month
  Pain will be recorded and graded using a 4-point scale (none, mild, moderate, or severe).

SECONDARY OUTCOMES:
Score on pain due to injection of rocuronium | 1 month
  Withdrawal reactions are scored as follows: (a) no pain response, (b)pain limited to the wrist, (c) pain limited to the elbow/shoulder, or (d) generalized pain response.

OTHER OUTCOMES:
To assess patient satisfaction | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Fakelma 05327079113, Principal Investigator — Diskapi Teaching and Research Hospital
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Altindag, Turkey (Türkiye)